CLINICAL TRIAL: NCT02552914
Title: Evaluation of the Use of the Colli-Pee Device to Collect First-void Urine for Molecular Detection of Several Sexual Transmitted Infections, Including Reproducibility of the Test Results and Acceptability by MSM Participating in a PrEP Study
Brief Title: Evaluation of the Use of the Colli-Pee Device to Collect First-void Urine for Molecular Detection of STIs
Acronym: Colli-Pee
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Novosanis NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 1027/15
Record Dates: First submitted 2015-08-28; First posted 2015-09-17 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Sexually Transmitted Diseases, Bacterial
Keywords: Colli-Pee; STI; first-void urine
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — First-void urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Colli-Pee — Participants will be asked to use the colli-pee to collect first-void urine and to send it back to the Institute of Tropical Medicine by regular mail.

SUMMARY:
Study objectives:

* To evaluate the usability of the Colli-PeeTM device to collect first-void urine for nucleic acid detection of Neisseria gonorrhoeae, Chlamydia trachomatis, Trichomonas vaginalis and Mycoplasma genitalium.
* To collect feedback on the easiness of use and the willingness of future use of the Colli-PeeTM device.

DETAILED DESCRIPTION:
Study population:

The Colli-Pee study is a sub-study of the Be-PrEP-ared study (EudraCT number: 2015-000054-37). All participants who participate in the Be-PrEP-ared study will be asked to participate in this sub-study.

Study design:

Participants who agree to be included in this study will be asked to collect first-void urine using the Colli-PeeTM device the day after the baseline, month 6, month 12 and month 18 visit. They will be asked to send the urine container back to ITM using regular mail. In addition they will also be asked to complete a small questionnaire concerning the easiness of use and the willingness of future use of the Colli-PeeTM device at the enrolment visit and final visit of the Be-PrEP-ared study.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the Be-PrEP-ared study
* Willing to collect first-void urine the next day and to send it back to ITM using regular mail.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only participants participating in the Be-PrEP-ared study (EudraCT number: 2015-000054-37) can be enrolled. These are men having sex with men who are at high risk acquiring HIV.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Detection of several STIs (CT/NG/MG/TV) on urine collected with the Colli-Pee device | up to 18 months
  To evaluate the use of the Colli-Pee device to collect first-void urine for nucleic acid detection of Neisseria gonorrhoeae, Chlamydia trachomatis, Trichomonas vaginalis and Mycoplasma genitalium.

SECONDARY OUTCOMES:
Easiness of use of the Colli-Pee device | up to 18 months
  Using a questionnaire the easiness of use of the Colli-Pee device will be assessed
Willingness of future use of the Colli-Pee device | up to 18 months
  Using a questionnaire the willingness of future use of the Colli-Pee device will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

REFERENCES:
- [Derived] De Baetselier I, Smet H, Abdellati S, De Deken B, Cuylaerts V, Reyniers T, Vuylsteke B, Crucitti T. Evaluation of the 'Colli-Pee', a first-void urine collection device for self-sampling at home for the detection of sexually transmitted infections, versus a routine clinic-based urine collection in a one-to-one comparison study design: efficacy and acceptability among MSM in Belgium. BMJ Open. 2019 Apr 3;9(4):e028145. doi: 10.1136/bmjopen-2018-028145. PMID 30948618